CLINICAL TRIAL: NCT06888830
Title: A Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Initial Efficacy of JS212 in Subjects With Advanced Malignant Solid Tumour
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JS212-001-I/II
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Advanced Malignant Solid Tumours
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS212 (Experimental): If needed, additional descriptive information (including which interventions are administered in each arm) to differentiate each arm from other arms in the clinical trial.
  Interventions: Drug: JS212 for Injection

INTERVENTIONS:
Drug: JS212 for Injection — JS212 for Injection is administered on the first day of the first cycle and every 3 weeks thereafter.

SUMMARY:
This study is a Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Initial Efficacy of JS212 in Subjects with Advanced Malignant Solid Tumour. Patients will be enrolled in two stages: a dose-escalation stage and a dose expansion stage.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of either sex who are 18 to 75 years of age (inclusive of 18 and 75 years) at the time of signing the consent form;
2. Histologically or cytologically confirmed advanced malignant solid tumors;
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
4. Expected survival of ≥ 12 weeks;
5. Subjects have at least 1 measurable lesion according to RECIST v1.1 criteria (without measurable lesions are allowed during dose escalation phase);

Exclusion Criteria:

1. Presence of active central nervous system metastasis. If previous radiotherapy or surgery, etc. has been received, and the imaging examination within 4 weeks before the first dose suggests that the brain metastasis is stable without exacerbation or new neurological symptoms, and hormone therapy has been discontinued two weeks before the first dose, screening is allowed; for the presence of meningeal metastasis and brainstem metastasis, regardless of the treatment or not, screening is not allowed;
2. Presence of clinically symptomatic pleural effusion, ascites, or pericardial effusion that requires repeated management (puncture or drainage, etc.);
3. Presence of medically uncontrolled hypertension, or with a history of hypertensive crisis or hypertensive encephalopathy;
4. Presence of a history of (non-infectious) interstitial lung disease (ILD)/non-infectious pneumonia requiring steroid therapy (e.g., idiopathic pulmonary fibrosis, mechanized pneumonia, drug-induced pneumonia, radiation pneumonitis, idiopathic pneumonia, etc.), and current ILD/non-infectious pneumonia;
5. Presence of clinically significant lung-specific co-morbidities including, but not limited to, any underlying lung disease (e.g., pulmonary embolism, severe asthma, severe COPD, restrictive lung disease, etc., diagnosed within 3 months prior to the first study dose) and any autoimmune, connective tissue, or inflammatory disease with pulmonary involvement (e.g., rheumatoid arthritis, Scheugelin's syndrome, sarcoidosis, etc.) and prior total pneumonectomy;
6. Presence of a history of immunodeficiency, including a positive test for Human Immunodeficiency Virus (HIV), or a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation；
7. the presence of other factors that may cause them to be forced to terminate the study midway, such as serious physical or mental illness or abnormal laboratory tests, which may increase the risk of participation in the study, affect treatment compliance, or interfere with the results of the study, and which, in the judgment of the investigator, make the subject unsuitable for participation in this study；

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
DLT | Up to 1 years
  Incidence and severity of DLT events
Incidence and severity of Adverse Events | Up to 2 years
  Abnormal changes in clinical symptoms, vital signs, physical examination, laboratory tests, electrocardiograph and other examinations.
MTD | Up to 1 years
  Maximum tolerated dose
RP2D | Up to 1 years
  Recommended phase II dose
ORR | Up to 2 years
  Objective Response Rate (ORR) as Assessed by Investigator according to RECIST v1.1

SECONDARY OUTCOMES:
DOR | Up to 2 years
  Duration of Objective Response (DOR) as Assessed by Investigator according to RECIST v1.1
DCR | Up to 2 years
  Investigator-assessed Duration of objective Response (DCR) according to RECIST v1.1
Progression-Free Survival (PFS) | Up to 2 years
  Progression-Free Survival (PFS) as Determined by Investigator according to RECIST v1.1
Overall Survival (OS) | Up to 2 years
  Overall Survival (OS)
Pharmacokinetic (PK) | About 6 months after first dosing
  Patient blood concentrations and pharmacokinetic parameters after drug administration
Immunogenicity | About 6 months after first dosing
  Incidence of antidrug antibodies (ADA)

OTHER OUTCOMES:
To explore the correlation between potential MARKERS and efficacy | Up to 2 years
  To explore the correlation between potential MARKERS and efficacy
To explore the correlation between serum β-Glucuronidase Concentrations and efficacy | Up to 2 years
  To explore the correlation between serum β-Glucuronidase Concentrations and efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No